CLINICAL TRIAL: NCT05584033
Title: Searching of Apraxia of Speech in Children With Specific Language Impairment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Samah Helmy Mohamed, residant, Sohag University
Other Study IDs: soh-med-22-10-09
Record Dates: First submitted 2022-10-12; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Apraxia of Speech
MeSH Terms: conditions — Apraxias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Mansora Arabic test battery for childhood apraxia of speech — Searching of apraxia of speech in children with Specific Language Impairment in able to better management of these cases.

SUMMARY:
Searching of Apraxia of Speech in Children with Specific Language Impairment

ELIGIBILITY:
Inclusion Criteria:

* Children from 4 to 8 years old diagnosed as specific language impairment

Exclusion Criteria:

* 1. Children with mental retardation or hearing impaired . 2. Children with any neurological or psychiatric disorders.

Ages: 4 Years to 8 Years | Sex: All
Age Groups: Child
Study Population: Searching of Apraxia of Speech in Children with Specific Language Impairment
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Mansora Arabic test battery for childhood apraxia of speech | one houre

CONTACTS AND LOCATIONS:
Locations (1):
- Sohage University, Sohage, Egypt